CLINICAL TRIAL: NCT06038305
Title: Prevalence of Anemia and Growth Assessment of Children Admitted With Acute Gastroenteritis in Assiut University Children Hospital
Brief Title: Prevalence of Anemia and Growth Assessment in Acute Gastroenteritis
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehad Ali Sayed, Resident physician, Family Medicine department, Assiut University
Other Study IDs: anemia and growth in AGE
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Acute Gastroenteritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Assessment of the growth parameters in infants admitted with acute gastroenteritis.
2. Determine the prevalence of anemia in infants admitted with acute gastroenteritis.

DETAILED DESCRIPTION:
Gastroenteritis is inflammation of the stomach, small intestine, or large intestine, leading to a combination of abdominal pain, cramping, nausea, vomiting, and diarrhea. Acute gastroenteritis usually lasts fewer than 14 days. Worldwide, gastroenteritis affects 3 to 5 billion children each year. Up to 40% of children aged less than 5 years with diarrhea are hospitalized with rotavirus. Also, some microorganisms have been found predominantly in resource-constrained nations, including Shigella spp, Vibrio cholerae, and the protozoan infections. Malnutrition, immunosuppression, young age, and an increase in the preceding diarrhea burdens are risk factors for the development of persistent diarrhea. A substantial proportion of global malnutrition is due to impaired intestinal absorptive function resulting from multiple and repeated enteric infections. These include recurrent acute infections as well as persistent infections, even those without overt liquid diarrhea.

Child growth is internationally recognized as the best global indicator of physical well-being in children because poor feeding practices-both in quantity and quality-and infections, or more often a combination of the two, are major factors that affect physical growth and mental development in children. The most important measurements needed for growth assessment are recumbent length or height, weight and head circumference. These fundamental anthropometric measures should be obtained and interpreted at each well child visit, and are typically sufficient for growth assessment.

In this study, the prevalence of anemia and growth of infants admitted with acute gastroenteritis at Assiut University Children Hospital will be assessed. Anemia is a global public health problem, with important consequences for human health and the social and economic development of each nation. It results from single or multiple causes that act simultaneously, influencing children's health, their cognitive and physical development, and immunity, increasing the risk of infections and infant mortality.

ELIGIBILITY:
Inclusion Criteria:

* Infants with acute gastroenteritis.
* Infants aged from 1 month and up to 2 years.

Exclusion Criteria:

* Infants aged less than 1 month and more than 2 years.
* Infants with persistent and chronic diarrhea.
* Infants with acute gastroenteritis in association with chronic disease

Ages: 1 Month to 2 Years | Sex: All
Age Groups: Child
Study Population: infants aged 1 month up to 2 years with acute gastroenteritis
Sampling Method: Non-Probability Sample
Enrollment: 297 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Determine association between anemia and acute gastroenteritis in infants and children. | baseline
  assess anemia in children with acute gastroenteritis and if anemia affect severity of acute gastroenteritis

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt